CLINICAL TRIAL: NCT01162382
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Major Depressive Disorder: A Functional Connectivity Magnetic Resonance Imaging (fcMRI) Study
Brief Title: Repetitive Transcranial Magnetic Stimulation for Treating Depression: A Functional Magnetic Resonance Imaging Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant support ended following which the key personnel (PI) left the institution.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WUSM3621222-201110079
Record Dates: First submitted 2009-11-30; First posted 2010-07-14 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder
Keywords: transcranial magnetic stimulation; TMS; rTMS; depression; fcMRI; EEG
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): Open-label transcranial magnetic stimulation
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Four 100-second trains and then one 65-second train, with 30-second inter-train intervals, at 1 Hz and 120% of the resting motor threshold will be applied over the right dorsolateral prefrontal cortex. Subsequently, twenty-five 30-second trains, with a 30-second inter-train interval, at 10 Hz and 120% of the resting motor threshold will be applied over the left dorsolateral prefrontal cortex.
  Other Names: Magstim Rapid stimulator

SUMMARY:
This protocol, "Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Major Depressive Disorder (MDD): A Functional Connectivity Magnetic Resonance Imaging (fcMRI) Study," is an open-label pilot treatment study. The purpose of the present protocol is to treat participants with a diagnosis of Major Depressive Disorder with 4 weeks of rTMS, performing fcMRI and EEG studies prior to and following treatment to determine if treatment response is related to changes in fcMRI and/or EEG results. The investigators hypothesize that patients who respond to treatment will display changes in functional connectivity patterns thought to be related to the occurrence of depressive symptoms.

DETAILED DESCRIPTION:
Depression is accompanied by rumination that supports inwardly focused cognitive attention on negative events and emotions. There is evidence to indicate that one aspect of this ruminative behavior lies in an abnormal increase in intra-regional connectivity among elements of the default mode network (DMN). It is also widely recognized that depression is associated with disturbances of cognition that include deficits in attentional processing, including both reductions in processing speed and deficits in selective attentional processing that are considered a part of executive function. Thus, there is at least equal reason to believe that attention and executive control networks might show changes in intra-regional functional connectivity. Given the attentional deficits associated with MDD, we hypothesize that there will be a weakening of intra-network resting state BOLD functional connectivity (rs-fcMRI) in addition to the strengthened connectivity reported by others.Further, we suggest that these shifts in intra-regional connectivity extend to the well-recognized anti-correlated activity between these two networks and support the intrusion of introspective, ruminative thought on cognitive activities that require externally directed attention. To test this hypothesis, we will use fMRI resting state functional connectivity to examine shifts in network connectivity prior to and following rTMS treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

SCREENING/DIAGNOSTIC REQUIREMENTS:

* Male or female outpatients, ages 18-50 (some literature has shown increasing cortical distance with age that may affect treatment outcome
* Hamilton Rating Scale of Depression (HRSD-24) > 18
* New onset major depression or untreated recurrent major depression per DSM-IV-TR38 criteria.
* Not taking antidepressant medication or any other psychotropic medication
* Using an adequate contraceptive method
* Able to give informed consent
* Available for 4 weeks of daily therapy, working hours, Mon.-Fri.
* English-speaking

Exclusion Criteria:

DIAGNOSTIC EXCLUSIONS:

* Co-morbid psychiatric diagnosis of bipolar disorder, acute OCD, schizophrenia or schizoaffective or concurrent treatment with outpatient ECT, or personality disorder or MDD with suicidal ideation as determined by history and/or by P.I. examination requiring hospital admission or referral for acute care.
* Previous failure to respond to treatment with rTMS
* Failure to achieve satisfactory improvement in depression after two or more adequate trials of antidepressant medications.

MEDICAL EXCLUSIONS:

* Patients newly diagnosed with thyroid dysfunction
* History of drug and/or ETOH dependence
* History of seizures
* History of head injury with loss of consciousness > 5 minutes
* Any implantable metal object in the skull or near their head
* Any implantable devices such as a cardiac pacemaker, vagal nerve stimulator, etc.
* Positive urine pregnancy test
* Severe migraine headaches uncontrolled with routine non-narcotic medication
* Any medical condition in the opinion of the Investigator that might confound the results of the study Contraindications to fcMRI procedure
* Intake of NSAIDS, narcotic or muscle relaxants within 72 hours of the fMRI protocol.
* Claustrophobia.
* Left-handedness (may influence cerebral cortical hemispheric dominance).
* Inability to tolerate, or medical contraindication to MRI testing (e.g. metal prostheses or implants, history of claustrophobia)

PROTOCOL SPECIFIC EXCLUSIONS:

* Unable to determine motor threshold for determining treatment dose with rTMS device
* Mini Mental Status Exam (MMSE)70 score < 24.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Garcia, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Demitrack MA, Thase ME. Clinical significance of transcranial magnetic stimulation (TMS) in the treatment of pharmacoresistant depression: synthesis of recent data. Psychopharmacol Bull. 2009;42(2):5-38. PMID 19629020
- [Background] Broyd SJ, Demanuele C, Debener S, Helps SK, James CJ, Sonuga-Barke EJ. Default-mode brain dysfunction in mental disorders: a systematic review. Neurosci Biobehav Rev. 2009 Mar;33(3):279-96. doi: 10.1016/j.neubiorev.2008.09.002. Epub 2008 Sep 9. PMID 18824195
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Savitz JB, Drevets WC. Imaging phenotypes of major depressive disorder: genetic correlates. Neuroscience. 2009 Nov 24;164(1):300-30. doi: 10.1016/j.neuroscience.2009.03.082. Epub 2009 Apr 7. PMID 19358877
- [Background] Zou K, Deng W, Li T, Zhang B, Jiang L, Huang C, Sun X, Sun X. Changes of brain morphometry in first-episode, drug-naive, non-late-life adult patients with major depression: an optimized voxel-based morphometry study. Biol Psychiatry. 2010 Jan 15;67(2):186-8. doi: 10.1016/j.biopsych.2009.09.014. PMID 19897176

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation
Started (No data are available fo this study as the study was terminated and PI has left the institution.) | 0
Completed (No data are available fo this study as the study was terminated and PI has left the institution.) | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No data are available for this study as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale-24 Point Version (HDRS-24)
Description: HDRS-24 will be used to measure response to rTMS treatment. A 50% decrease in HDRS-24 score will indicate treatment response; HDRS-24 < 10 will indicate remission.
Time Frame: At study entry and within 2 days of exiting 4 weeks of rTMS treatment
Population: as for baseline characteristics
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0

2. Secondary Outcome: fCMRI Results
Description: Imaging studies will be compared to determine if any changes in functional connectivity can be correlated with treatment response.
Time Frame: At study entry and within 2 days of exiting 4 weeks of rTMS treatment
Population: as for baseline characteristics
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No data are available for this study as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.
Description: No data are available for this study as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.
Arm/Group | Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No data are available for this study as the study was terminated and PI has left the institution. Multiple efforts to contact the PI for the relevant data have failed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No